CLINICAL TRIAL: NCT02871310
Title: Randomized, Double-Blind, Placebo-Controlled, Monocenter, Crossover Investigation to Evaluate the Vasoactive Effects of IQP-AS-118 in Healthy Individuals: A Pilot Study
Brief Title: Vasoactive Effects of IQP-AS-118 in Healthy Individuals
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study discontinued
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: INQ/030815
Record Dates: First submitted 2016-08-10; First posted 2016-08-18 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2018-01

CONDITIONS: Blood Flow; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IQP-AS-118 (Experimental): To be taken once daily dosing of 1 tablet in the morning with 250 mL of water. The tablets should not be chewed, but swallowed whole.
  Interventions: Dietary Supplement: IQP-AS-118
- Placebo (Placebo Comparator): To be taken once daily dosing of 1 tablet in the morning with 250 mL of water. The tablets should not be chewed, but swallowed whole.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: IQP-AS-118 — 1 tablet in the morning
  Arms: IQP-AS-118
Dietary Supplement: Placebo — 1 tablet in the morning
  Arms: Placebo

SUMMARY:
The main objective of this study is to evaluate the benefit of IQP-AS-118 on the vasoactive effects in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian males and females 45-65 years of age
2. Body mass index (BMI) of 25.0-29.9 kg/m2
3. Blood pressure (BP) at screening:

   * systolic blood pressure (SBP) ≤ 140 mmHg or
   * diastolic blood pressure (DBP) ≤ 90 mmHg
4. EndoPAT score: ≤ 2.00) at screening
5. Generally in good health, in particular an electrocardiogram (ECG) without pathological findings at screening
6. Readiness to comply with study procedures, in particular:

   * Consumption of the investigational product (IP) / placebo according to investigator's advise
   * Maintaining the same level of physical activity and usual diet during the entire study
   * Accepting blood draws
   * Able to undergo an EndoPAT assessment
   * Complying with visits and all respective requirements for BP and EndoPAT measurements
   * Filling in diaries/questionnaires
7. Non-smoker since at least 6 months prior to screening and during the study
8. Stable body weight in the last 3 months prior to screening (<3 kg self-reported change) and during the study
9. Concomitant medications must have been stable at least during the last 1 month prior to screening, if applicable
10. In women: postmenopausal for at least 12 months Participation is based upon written informed consent form (ICF) by the participant following written and oral information by the investigator regarding nature, purpose, consequences and possible risks of the clinical study.

Exclusion Criteria:

1. Known sensitivity to any components of the IP
2. Known primary or secondary hypertension or white-coat hypertension
3. Known impaired endothelial function as per investigator's judgement
4. Clinically significant disturbances in lipid metabolism e.g. known genetic hyperlipidemia
5. Known type-1 / type-2-diabetes
6. Untreated or non-stabilized thyroid disorder
7. History and/or presence of clinically significant cardiovascular disease as per investigator's judgement:

   1. Known congenital heart defects
   2. Myocardial infarction, heart failure, angina pectoris, life-threatening arrhythmia or stroke within the last 6 months prior to screening
   3. Existing thrombosis or disposition to thrombosis
8. Any other known significant or serious condition / disease that renders subjects ineligible, e.g.:

   1. History of malignancy within ≤5 years prior to screening
   2. Bleeding disorder and/or need for anticoagulants or anti-platelet agents
   3. Current psychiatric care and/or use of neuroleptics
   4. Bariatric surgery in the last 12 months prior to screening
9. Any known metabolic disease, gastrointestinal disorder or other clinically significant disease/disorder which in the investigator's opinion could interfere with the results of the study or the safety of the subject
10. Known arm lymphedema (e.g. due to mastectomy)
11. Other clinically relevant excursions of safety parameters or any other clinically significant abnormality in hematology and/or biochemistry at the Investigator's judgement
12. Dietary habits and/or restrictions that may affect the study outcome
13. Eating disorder or participation in a weight loss program
14. Use of medications (e.g. statins, renin angiotensin system inhibitors, nevibolol, carvedilol, calcium channel blockers) or supplements that can influence vascular endothelial function and/or blood flow (e.g. garlic, cocoa) within the last 4 weeks prior to screening and during the study
15. Use of antiplatelet agents and / or anticoagulants (e.g. warfarin, acetylsalicylic acid) within the last 4 weeks prior to screening and during the study
16. Use of medications or supplements that can influence SBP or DBP (e.g. ACE inhibitors, diuretics, calcium channel, α- or ß-blockers, grape seed extract, coenzyme Q10 etc.) within the last 4 weeks prior to screening and during the study
17. Use of lipid lowering medications (affecting lipid metabolism, platelet function or antioxidant status, etc.) and/or dietary supplements (e.g. omega-3 fatty acids, green tea extract, calcium, red yeast rice, phytosterols (incl. enriched products such as e.g. Becel), niacin,, glucomannan or chitosan ) within the last 4 weeks prior to screening and during the study
18. Use of medications that can influence cholesterol levels significantly (e.g. corticosteroids, amiodarone, estrogen, anabolic steroids) according to investigator's judgement
19. Use of weight loss treatment
20. Alcohol abuse (men: ≥21 units/week, women: ≥14 units/ week; 1 unit equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
21. Drug abuse
22. Reported participation in night shift work 2 weeks prior to screening and/or during the study
23. Participation in another study or blood donation during the last 30 days prior to screening and during the study
24. Any other reason deemed suitable for exclusion per investigator's judgment, e.g. insufficient compliance with study procedures

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in EndoPAT (chronic effect) | 12 weeks
  Pre-dose at the end vs. start of each intervention (week 4 vs. week 0 and week 12 vs. week 8, respectively) (inclusive of 4 weeks of wash-out period)

SECONDARY OUTCOMES:
Change in EndoPAT (acute effect) | 12 weeks
  3 h post-dose vs. pre-dose at start of each intervention (week 0 and week 8, respectively) (inclusive of 4 weeks of wash-out period)
Changes in ex vivo blood platelet aggregation / adhesion (acute effect) | 12 weeks
  3 h post-dose vs. pre-dose at start of each intervention (week 0 and week 8, respectively) (inclusive of 4 weeks of wash-out period)
Changes in ex vivo blood platelet aggregation / adhesion pre-dose (chronic effect) | 12 weeks
  End vs. start of each intervention (week 4 vs. week 0 and week 12 vs. week 8, respectively) (inclusive of 4 weeks of wash-out period)
Changes in blood coagulation / clotting parameters (acute effect) | 12 weeks
  3 h post-dose vs. pre-dose at start of each intervention (week 0 and week 8, respectively) (inclusive of 4 weeks of wash-out period)
Changes in blood coagulation / clotting parameters predose (chronic effect) | 12 weeks
  End vs. start of each intervention (week 4 vs. week 0 and week 12 vs. week 8, respectively) (inclusive of 4 weeks of wash-out period)
Global evaluation of benefit | 12 weeks
  Assessed by the subjects and investigator at end of each intervention (inclusive of 4 weeks of wash-out period)
Changes in SF- 12 | 12 weeks
  End vs. start of each intervention (week 4 vs. week 0 and week 12 vs. week 8, respectively) (inclusive of 4 weeks of wash-out period)
Physical examination | 12 weeks
  End of each intervention vs. screening (Week 4 vs. screening, week 12 vs. screening) (inclusive of 4 weeks of wash-out period)
Pulse rate | 12 weeks
  End vs. start of each intervention (Week 4 vs. week 0, week 12 vs. week 8) (inclusive of 4 weeks of wash-out period)
Systolic Blood Pressure | 12 weeks
  End vs. start of each intervention (Week 4 vs. week 0, week 12 vs. week 8) (inclusive of 4 weeks of wash-out period)
Diastolic Blood Pressure | 12 weeks
  End vs. start of each intervention (Week 4 vs. week 0, week 12 vs. week 8) (inclusive of 4 weeks of wash-out period)
Assessment of Adverse Events | 12 weeks
  Start and end of each intervention (Week 0, week 4, week 8 and week 12) (inclusive of 4 weeks of wash-out period)
Global assessment of tolerability | 12 weeks
  Assessed by the subjects and investigator (4-point categorical scale) at week 4 and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack, Principal Investigator — analyze & realize GmbH
Locations (1):
- analyze & realize GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No